CLINICAL TRIAL: NCT04308863
Title: Evaluation of Chitosan Scaffold and Mineral Trioxide Aggregate Pulpotomy in Mature Permanent Molars With Irreversible Pulpitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Instructor of Dental Public Health and Statistician, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chitosan vs MTA
Record Dates: First submitted 2020-03-09; First posted 2020-03-16 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Pulpitis - Irreversible

STUDY DESIGN:
Intervention Model Description: Thirty permanent mandibular molars of patients with signs and symptoms of irreversible pulpitis will be selected. They will be randomly allocated into two groups, Group 1(Chitosan scaffold/ MTA pulp dressing materials), Group 2 (MTA pulp dressing material).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chitosan scaffold/ MTA pulp dressing material (Experimental)
  Interventions: Drug: Chitosan scaffold/ MTA pulp dressing material
- MTA pulp dressing material (Active Comparator)
  Interventions: Drug: MTA pulp dressing material

INTERVENTIONS:
Drug: Chitosan scaffold/ MTA pulp dressing material — Chitosan 3-D porous scaffold will be prepared. The chitosan scaffolds will be examined with the Scanning electron microscopy (SEM) to analyze the surface of the chitosan scaffolds. The scaffolds will be sterilized by Ethylene oxide and stored until further use. A piece of 2-mm thick chitosan scaffold will be gently placed onto the pulp chamber floor and covering the canal orifices, and then a 2-3 mm thick layer of fast setting EndoCem Zr MTA will be applied onto the chitosan scaffold and will be gently condensed with moistened cotton pellet to attain adequate thickness which will be confirmed radiographically. MTA will be allowed to set for 4-5 mins.
  Arms: Chitosan scaffold/ MTA pulp dressing material
Drug: MTA pulp dressing material — MTA will be gently placed over the fresh pulp wound using an MTA carrier to a thickness of 2-3 mm. It will be condensed lightly with moistened cotton pellet to attain adequate thickness and confirmed radiographically. MTA will be allowed to set for 4-5 mins.
  Arms: MTA pulp dressing material

SUMMARY:
The aim of this study is to evaluate the clinical and radiographic outcomes of Chitosan scaffold and Mineral trioxide aggregate (MTA) when used as pulpotomy agents in mature permanent teeth with irreversible pulpitis.

DETAILED DESCRIPTION:
Thirty permanent mandibular molars of patients with signs and symptoms of irreversible pulpitis will be selected. They will be randomly allocated into two groups, Group 1(Chitosan scaffold/ MTA pulp dressing materials), Group 2 (MTA pulp dressing material). A single visit full pulpotomy procedure will be carried out. Chitosan scaffold and / or MTA will be used as the pulp dressing materials. The teeth will be then restored with base of Glass ionomer cement followed by composite restoration.

ELIGIBILITY:
Inclusion Criteria:

* Participants free from any systemic disease.
* Deep caries in a permanent lower molar with mature roots.
* Probing pocket depth and mobility within normal limits.
* No signs of pulpal necrosis including sinus tract or swelling.
* Vital bleeding pulp tissue should be present in all canals after complete pulpotomy.
* The tooth is restorable.
* Clinical diagnosis of symptomatic irreversible pulpitis based on subjective and objective examinations:

  * Subjective examination: Patients complaining of intermittent or spontaneous pain or pain exacerbated by dramatic temperature changes especially to cold stimuli and lasting for a few seconds to several hours.
  * Objective examination:

    * Clinical examination: Teeth that will experience immediate, excruciatingly painful sensation as soon as the cold stimulus is placed on and which may last for a while even after the removal of the stimulus.
    * Radiographic examination: Preoperative radiographs will be taken using a paralleling device.
    * The periapical index developed by Orstavik et al. (1986)(35) will be used to score cases with periapical rarefaction during diagnosis and follow-up periods. It consists of five categories:

      1. Normal periapical structures.
      2. Small changes in bone structures.
      3. Change in bone structure with mineral loss.
      4. Periodontitis with well-defined radiolucent area.
      5. Severe periodontitis with exacerbating features. Score 1 and 2 are considered healthy, score 3-5 are considered diseased
    * The teeth that will be included should have score 1 or 2.

Exclusion Criteria:

* Negative response to cold testing.
* No pulp exposure after caries excavation.
* Bleeding could not be controlled in 10 minutes after 2.5% NaOCl
* Absence of bleeding from any of the canals.
* Teeth with radiographic signs of internal resorption.
* Pulpal calcifications.
* Participants with stainless-steel wires and brackets.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | one week
  Postoperative pain will be recorded on Numerical Rating Pain Scale (NRS) that will be given to the patient to record his pain intensity in the range between 0-10, until the seventh day after treatment. Pain on the NRS will be further categorized as: No pain (0), Mild (1-3), Moderate (4-6), and Severe (7-10) pain.
Mineralization Activity | baseline
  Post-operative digital radio-graphic follow up will be done using the paralleling device to assess the rate of tooth mineralization
Mineralization Activity | 1 month
  Post-operative digital radio-graphic follow up will be done using the paralleling device to assess the rate of tooth mineralization
Mineralization Activity | 3 months
  Post-operative digital radio-graphic follow up will be done using the paralleling device to assess the rate of tooth mineralization
Mineralization Activity | 6 months
  Post-operative digital radio-graphic follow up will be done using the paralleling device to assess the rate of tooth mineralization
Mineralization Activity | 9 months
  Post-operative digital radio-graphic follow up will be done using the paralleling device to assess the rate of tooth mineralization
Mineralization Activity | 12 months
  Post-operative digital radio-graphic follow up will be done using the paralleling device to assess the rate of tooth mineralization
Root Canal Obliteration | baseline
  Post-operative digital radio-graphic follow up will be done using the paralleling device to assess the presence/absence of canal obliteration
Root Canal Obliteration | 1 month
  Post-operative digital radio-graphic follow up will be done using the paralleling device to assess the presence/absence of canal obliteration
Root Canal Obliteration | 3 months
  Post-operative digital radio-graphic follow up will be done using the paralleling device to assess the presence/absence of canal obliteration
Root Canal Obliteration | 6 months
  Post-operative digital radio-graphic follow up will be done using the paralleling device to assess the presence/absence of canal obliteration
Root Canal Obliteration | 9 months
  Post-operative digital radio-graphic follow up will be done using the paralleling device to assess the presence/absence of canal obliteration
Root Canal Obliteration | 12 months
  Post-operative digital radio-graphic follow up will be done using the paralleling device to assess the presence/absence of canal obliteration
Internal Root Resorption | baseline
  Post-operative digital radiographic follow up will be done using the paralleling device in order to assess the presence/absence of internal resorption
Internal Root Resorption | 1 month
  Post-operative digital radiographic follow up will be done using the paralleling device in order to assess the presence/absence of internal resorption
Internal Root Resorption | 3 months
  Post-operative digital radiographic follow up will be done using the paralleling device in order to assess the presence/absence of internal resorption
Internal Root Resorption | 6 months
  Post-operative digital radiographic follow up will be done using the paralleling device in order to assess the presence/absence of internal resorption
Internal Root Resorption | 9 months
  Post-operative digital radiographic follow up will be done using the paralleling device in order to assess the presence/absence of internal resorption
Internal Root Resorption | 12 months
  Post-operative digital radiographic follow up will be done using the paralleling device in order to assess the presence/absence of internal resorption

SECONDARY OUTCOMES:
Changes in the dental pulp in treated teeth | 6 months
  This will be performed in comparison to a non-affected tooth with clinical vitality and without any additional past treatment. All observers will analyze the images using the following rating scale regarding to alterations of signal intensity of the dental pulp at nT1w, fsT1w, and fsT2w at distinct time intervals (1 = no signs of alterations of signal intensity of the dental pulp between affected and non-affected teeth, 2 = slightly alterations of signal intensity of the dental pulp between affected and nonaffected teeth, and 3 = obvious alterations of signal intensity of the dental pulp between affected and nonaffected teeth)
Peri-radicular/furcal pathosis | 12 months
  Cone beam computed tomography (CBCT) analysis will be performed to detect presence/absence of any peri-radicular/furcal pathosis
Internal and external root resorption | 12 months
  Cone beam computed tomography (CBCT) analysis will be performed to detect presence/absence of internal or external root resorption

CONTACTS AND LOCATIONS:
Overall Officials: Maha T Aboul Kheir, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Rania M ElBackly, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Raef Sherif, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Yasser Elkamary, Study Chair — European Egyptian Pharmaceutical Industries, Pharco Corporation, Alexandria, Egypt; Nayera Mokhless, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Choukroun J, Diss A, Simonpieri A, Girard MO, Schoeffler C, Dohan SL, Dohan AJ, Mouhyi J, Dohan DM. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part IV: clinical effects on tissue healing. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e56-60. doi: 10.1016/j.tripleo.2005.07.011. PMID 16504852
- [Background] Parirokh M, Torabinejad M. Mineral trioxide aggregate: a comprehensive literature review--Part III: Clinical applications, drawbacks, and mechanism of action. J Endod. 2010 Mar;36(3):400-13. doi: 10.1016/j.joen.2009.09.009. PMID 20171353
- [Background] Kumar V, Juneja R, Duhan J, Sangwan P, Tewari S. Comparative evaluation of platelet-rich fibrin, mineral trioxide aggregate, and calcium hydroxide as pulpotomy agents in permanent molars with irreversible pulpitis: A randomized controlled trial. Contemp Clin Dent. 2016 Oct-Dec;7(4):512-518. doi: 10.4103/0976-237X.194107. PMID 27994420
- [Background] Li F, Liu X, Zhao S, Wu H, Xu HH. Porous chitosan bilayer membrane containing TGF-beta1 loaded microspheres for pulp capping and reparative dentin formation in a dog model. Dent Mater. 2014 Feb;30(2):172-81. doi: 10.1016/j.dental.2013.11.005. Epub 2013 Dec 12. PMID 24332410
- [Background] Ho MH, Kuo PY, Hsieh HJ, Hsien TY, Hou LT, Lai JY, Wang DM. Preparation of porous scaffolds by using freeze-extraction and freeze-gelation methods. Biomaterials. 2004 Jan;25(1):129-38. doi: 10.1016/s0142-9612(03)00483-6. PMID 14580916